CLINICAL TRIAL: NCT04125992
Title: Distal Radial Artery Access in Comparison to Forearm Radial Artery Access for Cardiac Catheterization, a Randomized Controlled Trial
Brief Title: Distal vs. Forearm Radial Artery Access
Acronym: DRAvsFRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: An-Najah National University (Other)
Responsible Party: Principal Investigator, Yunis Daralammouri, Assistant Professor, An-Najah National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRAvsFRA
Record Dates: First submitted 2019-09-29; First posted 2019-10-14 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Coronary Artery Disease; Angina, Unstable; Angina, Stable; Non STEMI; Non ST Segment Elevation Myocardial Infarction; Acute Coronary Syndrome; Atheroscleroses, Coronary; Atherosclerotic Heart Disease With Ischemic Chest Pain; Chest Pain; Myocardial Infarction; Myocardial Ischemia; ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: cardiac catheterization; coronary angiography; coronary angioplasty; snuff-box; snuffbox; snuff box; radial fossa; distal radial artery; radial artery; safeguard; distal radial access; distal radial angiography; radial access; angiography; distal radial; radial; coronary arteries; randomized controlled trial; left distal radial artery; Percutaneous Coronary Intervention; radial artery occlusion; forearm radial access; forearm radial artery; coronary catheterization; catheterization; left distal radial; angioplasty; coronary artery disease; radial vs distal
MeSH Terms: conditions — Coronary Artery Disease; Angina, Unstable; Angina, Stable; Non-ST Elevated Myocardial Infarction; Acute Coronary Syndrome; Chest Pain; Myocardial Infarction; Myocardial Ischemia; ST Elevation Myocardial Infarction; Arterial Occlusive Diseases | interventions — Angioplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patients enrolled to the study were randomized into Forearm Radial or Distal Radial groups. Care providers operated on patients and investigators collected their data during and after the operation. The independent variable - Access site (Forearm Radial or Distal Radial) - was coded into X or Z groups, then data was sent to the outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distal Radial (Experimental): Patients who undergo coronary catheterization by accessing the distal radial artery in the snuff-box of the hand.
  Interventions: Procedure: distal radial artery access in coronary angiography and angioplasty
- Forearm Radial (Active Comparator): Patients who undergo conventional coronary catheterization by accessing the forearm radial artery.
  Interventions: Procedure: Forearm radial artery access in coronary angiography and angioplasty

INTERVENTIONS:
Procedure: distal radial artery access in coronary angiography and angioplasty — The patient grasps his thumb towards the palm to bring the radial artery up to the surface. The left hand is set on the right side of the groin toward the operator, who stands on the right side, with the dorsal surface of hand upwards.
  Afterward, the access site is disinfected, lidocaine HCL is SC injected for local anesthesia. Subsequently, the distal radial artery is palpated to find the point of the strongest pulse. Later, at a 45-degree angle, the artery is punctured with a 21-gauge needle and a 0.018 soft, flexible, metallic wire is then inserted in the needle. Through the sheath, 200 micrograms of Nitroglycerin is given. A 5000 unit of unfractionated heparin is administered through the IV line. A weight-adjusted dose of heparin is further added if PCI is needed. Then, a 0.035 wire is introduced in the sheath with other required instruments such as the intracoronary device and the catheters. After pulling out the sheath, a compression device, Safe Guard, is used for hemostasis.
  Arms: Distal Radial
Procedure: Forearm radial artery access in coronary angiography and angioplasty — The right hand is set in the anatomical position, with the anterior surface of arm face upwards.
  Afterward, the access site is disinfected, lidocaine HCL is SC injected for local anesthesia. Subsequently, the forearm radial artery is palpated to find the point of the strongest pulse. Later, at a 45-degree angle, the artery is punctured with a 21-gauge needle and a 0.018 soft, flexible, metallic wire is then inserted in the needle. Through the sheath, 200 micrograms of Nitroglycerin is given. A 5000 unit of unfractionated heparin is administered through the IV line. A weight-adjusted dose of heparin is further added if PCI is needed. Then, a 0.035 wire is introduced in the sheath with other required instruments such as the intracoronary device and the catheters. After pulling out the sheath, a compression device, TR band, is used for hemostasis.
  Arms: Forearm Radial

SUMMARY:
The Distal Radial Access (DRA) to the coronaries has emerged recently. It's done via the distal radial artery in the radial fossa, which is known as the snuff-box. The rationale of conducting this research is to assess this new access advantages and disadvantages, in comparison with the standard conventional forearm radial access and examine if it's worthy to be a future alternative method for coronary angiography. It aims to randomly compare between the new distal radial access via the snuffbox and the conventional forearm radial access for percutaneous coronary angiography and angioplasty procedures. The objectives of comparing both procedures are to analyze the frequency of complications in terms of occlusion, arterial spasm, hematoma, and to weigh accesses effectiveness in terms of time and attempts to puncture, crossover rate, procedure duration, hemostasis time, and convenience of the patients and operators.

Candidates for coronary angiography are being randomized into the interventional group to undergo the angiography through the distal radial artery as the access site, or the control group accessing through the radial artery in the forearm. Procedural and post procedural outcomes and complications are being reported while patients are in hospital. All patients undergo doppler ultrasonography within 24 hours after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate in the study and sign the consent form.
* Patients with an indication for coronary catheterization
* Clinically stable patients
* Patients with palpable pulses on both access sites of the radial artery.

Exclusion Criteria:

* Patients with STEMI
* Patients with radial AV shunt for hemodialysis
* Patients with previous CABG using radial artery
* Patients with previous CABG using LIMA, RIMA or both.
* Patients with Renaud phenomenon or lymphedema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Radial artery occlusion | Within 24 hours after the procedure.
  Doppler Ultrasonography of the radial artery for occlusions along its course, in both groups.

SECONDARY OUTCOMES:
Puncture Time | During the procedure
  Which is time from first attempt to puncture to the successful one in seconds
Puncture Attempts | During the procedure
  Which is the number of puncture attempts from first one until the successful one (maximum 6)
Procedure Duration | During the procedure
  In minutes from the insertion of the sheath to its exertion.
Radiation Duration | During the procedure
  Which is measured by the radiological device in minutes.
Radiology Dose | During the procedure
  Which is measured by the radiological device in mGy.
Compression "hemostasis" time | Up to 240 minutes after band placement
  The time from the placement of the compression band until its removal (when there's no blood oozing after deflation), measured by minutes.
Arterial spasm | During the procedure
  Which is assessed by the operator if present or absent in terms of the difficulty in inserting the wire at the time of the procedures.
  of the procedure.
Hematoma and bleeding complications | Within 24 hours after the procedure
  It is defined by EASY hematoma scale.
Ischemic changes to the hand | Within 24 hours after the procedure
  It is noted by clinical features of pallor, absence of pulse, pain, cold, paresthesia or paralysis.
Crossover (failure to puncture) | During the procedure
  It is transforming from the selected access to another after 6 failed attempts to puncture the first selected access
Procedural pain | During the procedure
  Assessed by numerical rating scale (NRS) for pain, which is an 10 point subjective scale (0-10) where 0 refers for no pain, 1-3 for mild pain, 4-6 for moderate pain and 7-10 for severe pain.
Post-procedural pain | Within 24 hours after the procedure
  Assessed by numerical rating scale (NRS) for pain, which is an 11 point subjective scale (0-10) where 0 refers for no pain, 1-3 for mild pain, 4-6 for moderate pain and 7-10 for severe pain.
Rare complications | Within 24 hours after the procedure
  Pseudo-aneurysm, AV fistula formation, radial artery dissection, which are assessed by Doppler US. In addition to radial artery eversion or perforation.
Radial Artery Occlusion on follow up | After 2 weeks of the procedure.
  Follow up Doppler Ultrasonography for patients with occluded radial artery within 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Yunis Daralammouri, asst. prof., Principal Investigator — An-Najah National University
Locations (1):
- An-Najah National University Hospital, Nablus, Palestinian Territories